CLINICAL TRIAL: NCT07170644
Title: A Single-arm, Open-label Phase 2 Study of Nirogacestat in Adult Japanese Patients With Progressing Desmoid Tumors/Aggressive Fibromatosis (DT/AF)
Brief Title: A Study of Nirogacestat in Japanese Adults With Desmoid Tumors/Aggressive Fibromatosis (DT/AF)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: SpringWorks Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NIR-DT-202
Record Dates: First submitted 2025-07-31; First posted 2025-09-12 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Desmoid Tumor; Aggressive Fibromatosis
Keywords: Nirogacestat; PF-03084014; GSI; gamma secretase inhibitor; notch pathway; Ogsiveo
MeSH Terms: conditions — Desmoid Tumors | interventions — nirogacestat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nirogacestat (Experimental): Nirogacestat 150 mg by mouth, twice daily
  Interventions: Drug: Nirogacestat oral tablet

INTERVENTIONS:
Drug: Nirogacestat oral tablet — Nirogacestat tablet
  Other Names: PF-03084014; Ogsiveo

SUMMARY:
This study is being conducted to characterize the efficacy and safety of nirogacestat in Japanese adults with progressing desmoid tumors/aggressive fibromatosis.

DETAILED DESCRIPTION:
Desmoid tumors, also referred to as aggressive fibromatosis, are rare, locally invasive, slow growing soft tissue tumors. Although considered benign because of their inability to metastasize, desmoid tumors can cause significant morbidity and occasionally mortality in patients.

Nirogacestat is a tumor inhibitor that works by slowing or stopping the growth of tumor cells. Nirogacestat is a tablet taken by mouth and has been approved in the USA for adult patients with progressing desmoid tumors who require systemic treatment.

This is an open-label study to characterize the efficacy and safety of nirogacestat in Japanese adults with progressing desmoid tumors/aggressive fibromatosis (DT).

ELIGIBILITY:
Key Inclusion Criteria:

* Participant is aged ≥18 at the time of signing the informed consent.
* Participant has histologically confirmed DT (by local pathologist prior to informed consent) that has progressed by ≥20% as measured by RECIST v1.1 within 12 months of the screening visit scan.
* Participant has:

  1. Treatment-naive, measurably progressing DT that is deemed not amenable to surgery without the risk of significant morbidity; OR
  2. Recurrent, measurably progressing DT following at least 1 line of therapy; OR
  3. Refractory, measurably progressing DT following at least 1 line of therapy.
* Participant agreed to provide archival or new tumor tissue for re-confirmation of disease.
* Participant has a DT tumor where continued PD will not result in immediate significant risk to the participant.
* Participants who are receiving chronic NSAIDs as treatment for conditions other than DT must be receiving them prior to documented DT progressive disease (inclusion criterion 2) and on a stable dose for at least 28 days prior to the first dose of study treatment.
* Participant has an Eastern Cooperative Oncology Group (ECOG) performance status ≤2 at screening
* Participant has adequate organ and bone marrow function

Key Exclusion Criteria:

* Participant has known malabsorption syndrome or preexisting gastrointestinal conditions that may impair absorption of nirogacestat.
* Participant has experienced any of the following within 6 months of signing informed consent: clinically significant cardiac disease (New York Heart Association Class III or IV), myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass graft, symptomatic congestive heart failure, cerebrovascular accident, transient ischemic attack, or symptomatic pulmonary embolism.
* Participant has had lymphoma, leukemia, or any malignancy within the past 5 years at the time of informed consent, except for any locally recurring cancer that has been treated curatively (e.g., resected basal or squamous cell skin cancer, superficial bladder cancer, carcinoma in situ of the cervix or breast), with no evidence of metastatic disease for 3 years at the time of informed consent.
* Participant has known severe hepatic impairment
* Participant previously received or is currently receiving gamma secretase inhibitors or anti-Notch antibody therapy
* Participant is currently using any treatment for DT/AF including tyrosine kinase inhibitors (TKIs) or any investigational treatment 28 days (or 5 half-lives, whichever is longer) prior to the first dose of study treatment
* Participant is currently using or anticipates using food or drugs that are known strong/moderate cytochrome P450 (CYP) 3A4 inhibitors, or strong CYP3A inducers within 14 days prior to the first dose of study treatment.
* Participant has experienced other severe acute or chronic medical or psychiatric conditions within 1 year of signing informed consent.
* Participant is unable to comply with study related procedures (including, but not limited to, the completion of electronic patient-reported outcomes)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-08-08 (Actual); Primary Completion 2028-05-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | On the first day of every 3 cycles (each cycle is 28 days) until disease progression is observed or death, assessed up to approximately 3 years.
  Objective response rate (ORR), defined as the proportion of participants with confirmed complete response (CR) + partial response (PR) assessed by independent Central Imaging Review using RECIST v1.1 (Eisenhauer 2009).

SECONDARY OUTCOMES:
Duration of response (DoR) | On the first day of every 3 cycles (each cycle is 28 days) until disease progression is observed or death, assessed up to approximately 3 years.
  Duration of response (DoR), defined as the time from the first objective response (CR or PR) that is subsequently confirmed until the first occurrence of disease progression (radiographic or clinical) by RECIST v1.1 or death by any cause (whichever occurs first).
Time to Response (TTR) | On the first day of every 3 cycles (each cycle is 28 days) until disease progression is observed or death, assessed up to approximately 3 years.
  Time to Response (TTR), defined as the time interval between the first dose of study treatment and the first date of objective response that is subsequently confirmed.
Safety endpoints will include incidence of treatment-emergent adverse events (TEAEs), changes in laboratory parameters, vital signs, physical examination findings, and ECGs. | On the first day of every 3 cycles (each cycle is 28 days) until disease progression is observed or death, assessed up to approximately 5 years.
  Tolerability will be assessed according to toxicities graded by NCI CTCAE v5.0.
Progression Free Survival (PFS) | On the first day of every 3 cycles (each cycle is 28 days) until disease progression is observed or death, assessed up to approximately 3 years.
  Progression Free Survival (PFS) is defined as the time from the start of study treatment until the date of assessment of progression or death by any cause. Progression will be determined radiographically using RECIST v1.1 (Eisenhauer 2009) or clinically as assessed by the investigator.
  Clinical progression is defined as the onset or worsening of symptoms resulting in a global deterioration of health status causing the permanent discontinuation from study treatment and the initiation of emergent treatment (e.g., radiotherapy, surgery, or systemic therapy, including chemotherapy or tyrosine kinase inhibitors) for DT.
Symptoms and impacts will be assessed by evaluating change from baseline at Cycle 10 on the following patient reported outcomes (PROs): | On the first day of every 3 cycles (each cycle is 28 days) until disease progression is observed or death, assessed up to approximately 3 years.
  * Brief Pain Inventory (BPI) short form
  * European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire-Core 30 (QLQ-C30)
Characterize nirogacestat serum concentrations. | On the first day of the first cycle and of every third cycles (each cycle is 28 days) until disease progression is observed or death, assessed up to approximately 3 years.

CONTACTS AND LOCATIONS:
Locations (3):
- Japan (3):
  - Nagoya University Hospital, Nagoya, Aichi-ken
  - National Cancer Center Hospital, Chuo Ku, Tokyo
  - Osaka Prefectural Hospital Organization Osaka International Cancer Institute, Osaka

IPD SHARING:
Plan to Share IPD: Yes
SpringWorks Therapeutics is committed to data transparency and sharing data to further research while maintaining the privacy and confidentiality of research participants. Pertinent patient-level data from completed registrational clinical trials will be made available by SpringWorks to qualified researchers upon approval of reasonable requests following de-identification/anonymization pursuant to applicable law.